CLINICAL TRIAL: NCT05939375
Title: The Effect of Family-centered Care Educational Training on Nurses' Attitudes and Parental Satisfaction: A Semi-experimental Study
Brief Title: The Effect of Family-centered Care Educational Training on Nurses' Attitudes and Parental Satisfaction
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Derya AKDENIZ UYSAL, PhD, Nursing, Mersin University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: MersinU-HB-OGP-01
Record Dates: First submitted 2023-06-13; First posted 2023-07-11 (Actual); Last update posted 2023-07-11 (Actual); Status verified 2023-07

CONDITIONS: Nursing Care
Keywords: nursing; family centered care; attitute; satisfaction
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Intervention Model Description: This non-randomized experimental study, which employs a pre/post-test design, was conducted with the participation of 130 nurses and 100 parents. An educational training, grounded in six weeks of nurse centered interactions, was implemented. Nurse centered interactions and group discussions were conducted by supervising nurses with at least a master of science degree in pediatric nursing, together with the researchers. One week before the educational training, the nurses were administered the Nurse Information Form and FCCAS pre tests, which were conducted using an online form.Six weeks after the completion of the six week educational training, the nurses were administered the FCCAS post-test via an online form.The PedsQL HCPSS was utilized to assess the level of healthcare satisfaction among parents whose children received care in pediatric clinics.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FCC educational training (Experimental): The administration of the pre-tests, the planning of the educational process, including the development of e-learning modules and video lectures, was shared with the nurses.Each week, the topics were delivered to the nurses through online interactive methods, with each session lasting approximately 45-60 minutes. Six weeks after the completion of the six-week educational training, the nurses were administered the FCCAS post test via an online form.
  The PedsQL HCPSS was utilized to assess the level of healthcare satisfaction among parents whose children received care in pediatric clinics. To assess parental healthcare satisfaction before the training, the mean scores of the PedsQL HCPSS from the institutional data of the hospital in January 2021 were used. Post training parental data were collected in May-June 2021 using the PedsQL HCPSS from parents whose children received care in pediatric clinics.
  Interventions: Behavioral: FCC educational training

INTERVENTIONS:
Behavioral: FCC educational training — An educational training, grounded in six weeks of nurse-centered interactions, was implemented.

SUMMARY:
Family-Centered Care (FCC) is a care approach based on mutual respect, knowledge sharing, and collaboration among children, families, and healthcare professionals during the planning, implementation, and evaluation of healthcare. Nurses' supportive attitudes may positively influence their care practices and behaviors towards FCC. In this regard, educational training related to FCC may affect nurses' attitudes and behaviors. In the literature, it's evident that there is a need for studies examining how both the attitudes of nurses towards FCC a key determinant of their behavioral predispositions, and the parental satisfaction with healthcare services change in response to the provision of educational training. This study aims to determine the impact of the FCC educational training administered to nurses in pediatric clinics, primarily on nurses' attitudes towards FCC, and secondarily on parental satisfaction with healthcare. With this in mind, this study aims to determine the primary impact of the nurse centered FCC educational training, provided to nurses in pediatric clinics, on nurses' attitudes towards FCC, and its secondary impact on parental satisfaction with healthcare.

DETAILED DESCRIPTION:
Research Hypotheses H1: There is a difference between the mean scores of nurses' attitudes towards FCC before and after the educational training.

H2: There is a difference between the mean scores of parental satisfaction with healthcare before and after the educational training.

This study employs a non randomized experimental design with a pre test, post test format. It was conducted between February and June 2021 in the pediatric units of a university hospital in the Eastern Mediterranean region of Turkey. The target population comprised 134 nurses working across a variety of specializations including pediatric hematology, pediatric surgery, pediatric emergency care, pediatric intensive care (PICU), neonatal intensive care (NICU), pediatric infectious diseases, and general pediatrics. In this study, where specific sample selection was not applied, the aim was to reach at least 80% of the total population. The research was undertaken with the participation of 130 nurses, which accounted for 97% of the targeted population.

Data collection tools; Nurse Information Form: These questions pertain to the nurses' age, gender, education, length of professional experience, duration spent in pediatric clinics, and prior participation in FCC training.

Family Centered Care Attitude Scale (FCCAS): The measurement tool, developed by Kara and Güdücü Tüfekçi, is used to identify the attitudes of nurses providing care to children and their parents towards FCC. This self-report tool is composed of 58 Likert scale items distributed across two subscales. An increase in the scale score indicates an increase in positive attitudes of nurses towards FCC.

PedsQL Health Care Parents Satisfaction Scale (PedsQL HCPSS): The PedsQL Health Care Parents Satisfaction Scale, originally designed by Varni and later adapted for Turkish audiences by Ulus and Kublay, is a self-report instrument used for assessing the satisfaction levels of parents whose children are utilizing healthcare services. Comprising 25 items divided into six subscales. A higher score on this scale signifies increased satisfaction among parents with the provided healthcare services.

Interventions The planning of the educational intervention process, the development of e-learning modules, and the organization of nurse centered interactions benefited from expert opinions in three nursing education, ten pediatric nursing, and two educational sciences. A six week period February - April 2021 was planned for the educational training. One week before the educational training, the nurses were administered the Nurse Information Form and FCCAS pre tests, which were conducted using an online form. Immediately following the administration of the pre tests, the planning of the educational process, including the development of e-learning modules and video lectures, was shared with the nurses. Each week, the topics were delivered to the nurses through online interactive methods, with each session lasting approximately 45-60 minutes. Complementing these sessions, video lectures of around 30 minutes duration were prepared for each topic. The flexibility of the e-learning format allowed nurses to access these modules and video lectures from any location. From the second week of the educational training, nurse centered interactions and group discussions were initiated within the clinical setting, providing a platform for collaborative learning and engagement among the nurses. In this process, at the beginning of each shift, FCC practices for children and their parents were discussed. In intra team interactions, group discussions were to explore the content of each week's module. Six weeks after the completion of the six week educational training, the nurses were administered the FCCAS post test via an online form. The PedsQL HCPSS was utilized to assess the level of healthcare satisfaction among parents whose children received care in pediatric clinics.

Statistical Methods Data analysis was conducted using SPSS version 21 (Statistical Package for Social Sciences) software. The Kolmogorov-Smirnov test was utilized to assess the normal distribution of the scale scores. Descriptive statistics such as mean, standard deviation, confidence interval, frequency, percentage, and effect size (d) were used to present the data. Paired sample t tests were employed to compare the mean scores of the FCCAS before and after the training among the nurses. Furthermore, the mean scores of the PedsQL HCPSS in the post training period were compared to the pre training institutional data of the hospital using a one sample t test.

Ethical Considerations The study obtained approval from the clinical research ethics committee, written institutional permission from the hospital, and informed consent from both the participating nurses and parents.

ELIGIBILITY:
Inclusion Criteria:

For nurses:

1. be working in the pediatric clinics between February and April 2021,
2. be willing to participate in the research.

For parents:

1. have a child receiving healthcare in the specified pediatric clinics during the period of May to June 2021 (post-training period),
2. be willing to participate in the research.

Exclusion Criteria:

For nurses:

1. don't be working in the pediatric clinics between February and April 2021,
2. not willing to participate in the research.

For parents:

1. haven't a child receiving healthcare in the specified pediatric clinics during the period of May to June 2021 (post-training period),
2. not willing to participate in the research.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 134 (Actual)
Dates: Start 2021-02-20 (Actual); Primary Completion 2021-04-20 (Actual); Study Completion 2021-06-20 (Actual)

PRIMARY OUTCOMES:
pediatric nurses' attitudes | an average of 3 month
  FCC educational training administered to nurses in pediatric clinics, improving on nurses' attitudes towards FCC.Family Centered Care Attitude Scale (FCCAS): The measurement tool, developed by Kara and Güdücü Tüfekçi, is used to identify the attitudes of nurses providing care to children and their parents towards FCC. This self-report tool is composed of 58 Likert scale items distributed across two subscales. An increase in the scale score indicates an increase in positive attitudes of nurses towards FCC.

SECONDARY OUTCOMES:
satisfaction with healthcare | an average of 2 month
  increasing on parental satisfaction with healthcare. PedsQL Health Care Parents Satisfaction Scale (PedsQL HCPSS): The PedsQL Health Care Parents Satisfaction Scale, originally designed by Varni and later adapted for Turkish audiences by Ulus and Kublay, is a self-report instrument used for assessing the satisfaction levels of parents whose children are utilizing healthcare services. Comprising 25 items divided into six subscales. A higher score on this scale signifies increased satisfaction among parents with the provided healthcare services.

CONTACTS AND LOCATIONS:
Locations (1):
- Mersin University, Mersin, Turkey (Türkiye)

REFERENCES:
- See also: Rostami, F., Hassan, S. T. S., Yaghmai, F., Ismaeil, S. B., & BinSuandi, T. (2015). The effect of educational intervention on nurses' attitudes toward the importance of family-centered care in pediatric wards in Iran. Electronic physician, 7(5), 1261. — https://pubmed.ncbi.nlm.nih.gov/26435826/
- See also: Angelo, M., Cruz, A. C., Mekitarian, F. F. P., & Martins, M. et al. (2014). Nurses' attitudes regarding the importance of families in pediatric nursing care. Revista da Escola de Enfermagem da USP, 48 — https://pubmed.ncbi.nlm.nih.gov/25517838/
- See also: Boztepe, H., & Kerimoğlu-Yıldız, G. (2017). Nurses perceptions of barriers to implementing family-centered care in a pediatric setting: A qualitative study. Journal for Specialists in Pediatric Nursing, 22(2), e12175. — https://pubmed.ncbi.nlm.nih.gov/28198079/
- See also: Feeg, V. D., Paraszczuk, A. M., Çavuşoğlu, H., & Al Mamun, A. et al. (2016). How is family centered care perceived by healthcare providers from different countries? An international comparison study. Journal of Pediatric Nursing, 31(3), 26 — https://pubmed.ncbi.nlm.nih.gov/26712214/